CLINICAL TRIAL: NCT02135315
Title: One-year Outcome of Intensive Versus Standard Blood Pressure Treatment in Non-ST Elevation Acute Coronary Syndrome: A Randomised Controlled Trial
Brief Title: Intensive Arterial Pressure Control in Acute Coronary Syndrome
Acronym: IAPREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Collaborators: Emergency NGO Onlus (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IAPREC
Record Dates: First submitted 2014-03-27; First posted 2014-05-09 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome, arterial pressure
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Isosorbide Dinitrate

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The assessments of outcome is conducted by aninvestigator who did not participate in the randomization, protocol treatment or in-hospital clinical treatment of the patient.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intensive controle group (Experimental): The end point in this group was to maintain the systolic blood pressure (SBP) between 110 and 120 mmHg using continuous intravenous Isosorbide Dinitrate perfusion, and Labetalol if needed.
  Interventions: Drug: Isosorbide Dinitrate
- standard control group (Active Comparator): The end point in these group was to maintain the systolic blood pressure under 140 mmHg using continuous intravenous Isosorbide Dinitrate perfusion, and Labetalol if needed.
  Interventions: Drug: Isosorbide Dinitrate

INTERVENTIONS:
Drug: Isosorbide Dinitrate — administration of continuous intravenous isosorbide dinitrate to obtain a SBP between 110 and 120 mmHg. After 2 hours from the start of treatment and if the blood pressure goal is not achieved, labetalol is used
  Other Names: Risordan

SUMMARY:
The intensive arterial pressure control in acute coronary syndrome (ACS) during the first 24 hours can improve the prognosis in the short and long term.

the study compare two treatment strategies (standard and intensive treatment) to assess their efficacy and safety in the treatment of acute coronary syndrome.

DETAILED DESCRIPTION:
Acute coronary syndrome is often associated with arterial pressure elevation which are deleterious for the heart and needs urgent intervention to lower the blood pressure to the required values, however there is no clear recommendations concerning the treatment intensity in this situation.

The investigators know that high arterial pressure increases the oxygen myocardial consumption and it is deleterious in acute coronary syndrome, so , it is logical to reduce intensively this pressure.

ELIGIBILITY:
Inclusion Criteria:

* Non-ST segment elevation Acute Coronary Syndrome

Exclusion Criteria:

* SBP under 90 mmHg or hemodynamic instability
* Complicated ACS (arrythmias, atrio-ventricular block, shock, tamponade...) or ST elevation myocardial infarction (STEMI)
* Patients with contraindication to nitrates and/or beta blockers

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
mortality | 12 months
  1-year death rate
major cardiovascular events (MACE) | 12months
  1-year MACE rate
combined mortality and MACE rate | 1 year
  combined mortality and MACE rate at one year.

SECONDARY OUTCOMES:
troponin change | 24 hours after baseline measurement
  troponin change between baseline and 24 hour after
Adverse events | 24 hours after start of protocol intervention
  Severe hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, MD, Principal Investigator — University of Monastir
Locations (1):
- university of Monastir, Monastir, Tunisia

REFERENCES:
- See also: official department website — http://www.urgencemonastir.com